CLINICAL TRIAL: NCT06672068
Title: To Evaluate the Efficacy and Safety of TY-9591 Tablets Combined With Chemotherapy as First-line Treatment in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) Harboring EGFR Mutation
Brief Title: A Study of TY-9591 With Chemotherapy as 1st Line Treatment in Patients With Mutated Epidermal Growth Factor Receptor NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TYK Medicines, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TYKM1601203
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-11

CONDITIONS: NSCLC
MeSH Terms: interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): TY-9591 80mg QD+pemetrexed 500mg/m²（D1，Q3w）+Carboplatin AUC5/ Cisplatin 75mg/m²（D1，Q3w*4 cycles）
  Interventions: Drug: TY-9591 80mg QD+pemetrexed+Cisplatin/Carboplatin
- Cohort 2 (Experimental): TY-9591 160mg QD+pemetrexed 500mg/m²（D1，Q3w）+Carboplatin AUC5/ Cisplatin 75mg/m²（D1，Q3w*4 cycles）
  Interventions: Drug: TY-9591 160mg QD+pemetrexed+Cisplatin/Carboplatin

INTERVENTIONS:
Drug: TY-9591 80mg QD+pemetrexed+Cisplatin/Carboplatin — TY-9591 80mg QD+pemetrexed 500mg/m²（D1，Q3w）+Carboplatin AUC5/ Cisplatin 75mg/m²（D1，Q3w*4 cycles）
  Other Names: TY-9591 +pemetrexed+Cisplatin/Carboplatin
  Arms: Cohort 1
Drug: TY-9591 160mg QD+pemetrexed+Cisplatin/Carboplatin — TY-9591 160mg QD+pemetrexed 500mg/m²（D1，Q3w）+Carboplatin AUC5/ Cisplatin 75mg/m²（D1，Q3w*4 cycles）
  Other Names: TY-9591+pemetrexed+Cisplatin/Carboplatin
  Arms: Cohort 2

SUMMARY:
This study was a parallel, randomized, multicenter phase II clinical trial to evaluate the efficacy and safety of TY-9591 combined with platinum-based chemotherapy as first-line treatment in patients with locally advanced or metastatic non-small cell lung cancer harboring EGFR sensitive mutations.

DETAILED DESCRIPTION:
Participants were randomly assigned in a 1:1 ratio to either cohort 1 or cohort 2 for 21-day treatment cycles until disease progression (RECIST v1.1 criteria), treatment discontinuation criteria, withdrawal criteria, or study discontinuation, whichever occurred first. After the subjects terminate or withdraw from this study, the investigators can use reasonable follow-up treatment according to the subjects' condition.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years old and <80 years old.
2. Patients with non-squamous non-small cell lung cancer (NSCLC) diagnosed by histology or cytology as locally advanced (clinical stage IIIB, IIIC, no chance of radical surgery or radical chemoradiotherapy) or metastatic (clinical stage IVA, IVB) (according to the AJCC TNM staging criteria for lung cancer, 8th edition).
3. Tissue or blood samples tested positive for EGFR sensitive mutations (including exon 19 deletion, exon 21 L858R mutation, alone or in combination with other EGFR mutations) by central laboratory or research center, other tertiary hospitals, or third-party laboratories.
4. He had received no previous systemic antitumor therapy for locally advanced or metastatic non-small-cell lung cancer. Patients who had received previous adjuvant and neoadjuvant therapy and definitive radiotherapy/chemoradiotherapy were allowed if the last treatment was more than 12 months after disease recurrence or metastasis.
5. Patients had at least one measurable target lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1) : no previous local treatment such as radiotherapy, an accurately measurable target lesion at baseline, and a baseline maximum diameter of 10mm or more (or a short diameter of 15mm or more in the case of a lymph node). For patients with postoperative recurrence, lesions in the area of previous local treatment (radiotherapy or other therapy) were considered measurable only if disease progression occurred more than 6 months after the end of treatment.
6. With an ECOG score of 0-1 and no deterioration during the first 2 weeks of the study, survival was expected to be no less than 3 months.
7. Patients were required to have adequate bone marrow reserve and no hepatic, renal, or coagulopathy, with laboratory values that met the following criteria (no previous blood or platelet transfusion, albumin, recombinant human thrombopoietin, or colony-stimulating factor (CSF) transfusion within 14 days before the first dose in this study).
8. Male patients and female patients of reproductive age should take adequate contraceptive measures within 3 months after signing the study informed consent to the last study drug treatment; In women of childbearing age, the blood pregnancy test results were negative within 7 days before the first dose.
9. Before the first dose of study drug, all toxic effects (except alopecia and grade 2 neurotoxicity related to prior platinum-based chemotherapy) associated with previous systemic therapy (e.g., adjuvant chemotherapy) had been resolved (to grade 1 or less).

Exclusion Criteria:

1. The following treatments exist for patients:

   1. Previous treatment with any EGFR-TKI was performed.
   2. Previous systemic anti-tumor therapy for advanced/metastatic non-small cell lung cancer (including chemotherapy, targeted therapy, biological therapy, immunotherapy, etc.), neoadjuvant and adjuvant therapy, definitive radiotherapy/chemoradiotherapy were eligible according to the inclusion criteria
   3. Anti-tumor therapy with traditional Chinese medicine with anti-tumor indications was received within 7 days before the first dose of the study drug.
   4. Prior whole brain radiotherapy (WBRT); Received >30% bone marrow or extensive radiation within 28 days before the first dose of study drug; Local radiotherapy or palliative radiotherapy for bone metastases had been administered within 7 days before the first dose of study drug.
   5. Uncontrolled or poorly controlled pleural effusion and pericardial effusion.
2. Patients with other malignancies or a history of other malignancies were excluded if they had malignancies that had been treated with curative intent, had no known active disease for more than 5 years before the first dose of study treatment, and had a low potential risk of recurrence; Cured basal cell or squamous cell carcinoma of the skin, papillary carcinoma of the thyroid, carcinoma in situ of the cervix and ductal carcinoma in situ of the breast.
3. rimary malignant brain tumors or unstable brain metastases. Unstable brain metastases were defined as patients with CNS complications requiring urgent neurosurgical treatment (e.g., surgery); Patients requiring glucocorticoids, mannitol, or diuretics with a dose of more than 5mg dexamethasone equivalent for the control of symptoms of brain metastases within 14 days before the first dose; Patients who received local radiotherapy or gamma knife treatment or other local CNS treatment (e.g., intrathecal chemotherapy) within 14 days before the first study dose; Patients with meningeal metastases were not enrolled.
4. The patient had symptoms of spinal cord compression caused by the tumor.
5. Uncontrollable cancer pain; Stable doses of narcotic painkillers were not achieved at enrollment.
6. Clinically significant gastrointestinal abnormalities that may affect the intake, transport, or absorption of the study drug, such as inability to take drugs orally, uncontrollable nausea or vomiting, history of large gastrointestinal resection, Uncured recurrent diarrhea, atrophic gastritis (onset age less than 60 years), uncured gastric diseases requiring long-term use of ppis, Crohn's disease, and ulcerative colitis.
7. A previous or screening history of interstitial lung disease or interstitial pneumonia (ILD), or drug-induced ILD, or radiation pneumonitis requiring hormonal therapy, or the presence of any evidence of active ILD (e.g., acute onset or progressive pneumonitis/pulmonary fibrosis at baseline) Or pulmonary symptoms that were considered by the investigator to be ineligible for enrollment or factors that were judged to be at high risk for the development of interstitial lung disease.
8. Had previously received an allogeneic bone marrow transplant.
9. Pregnant and lactating women.
10. Known or suspected allergy to test drug ingredients or their analogues.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to 33 months
  Defined as the proportion of subjects with an optimal response of CR or PR observed throughout the study from the start of randomization until first disease progression

SECONDARY OUTCOMES:
PFS | Up to 45 months
  It was defined as the time from the start of randomization to the first occurrence of disease progression or death from any cause, whichever occurred first
DoR | Up to 45 months
  It was defined as the time during study treatment from the first assessment of a tumor as CR or PR to the first assessment of PD or death from any cause, whichever occurred first
DCR | Up to 33 months
  The optimal response observed throughout the study from randomization to first disease progression was the proportion of subjects with CR or PR or SD (duration ≥6 weeks)
OS | Up to 45 months
  It was defined as the time from the start of randomization to death from any cause

IPD SHARING:
Plan to Share IPD: No